CLINICAL TRIAL: NCT03332732
Title: VNRX-5133-103: A Randomized, Drug-Drug Interaction Study to Assess the Safety and Pharmacokinetics of VNRX-5133 in Healthy Adult Volunteers
Brief Title: VNRX-5133 Drug-Drug Interaction in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-5133-103; 272201300019C-3-0-1 (NIH); 17-0068 (Other: DMID)
Record Dates: First submitted 2017-09-28; First posted 2017-11-06 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Bacterial Infections
Keywords: Healthy Volunteers; Pharmacokinetics
MeSH Terms: conditions — Bacterial Infections | interventions — taniborbactam; Metronidazole

STUDY DESIGN:
Intervention Model Description: Part 1: Cross-over Part 2: Parallel
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A (Experimental): In Part 1A, subjects will receive single doses of VNRX-5133 and VNRX-5022 alone and in combination. All subjects will receive all treatments in the sequence specified by the randomization schedule..
  Interventions: Drug: VNRX-5133; Drug: VNRX-5022
- Part 1B (Experimental): In part 1B, subjects from Part 1A will receive metronidazole with or without VNRX-5133 + VNRX-5022. All subjects will receive all treatments in the sequence specified by the randomization schedule.
  Interventions: Drug: VNRX-5133; Drug: VNRX-5022; Drug: Metronidazole
- Part 2 - 2A (Experimental): Multiple dose administration of Low Dose VNRX-5133 + VNRX-5022
  Interventions: Drug: VNRX-5133; Drug: VNRX-5022
- Part 2 - 2B (Experimental): Multiple dose administration of High Dose VNRX-5133 + VNRX-5022
  Interventions: Drug: VNRX-5133; Drug: VNRX-5022
- Part 2 - 2C (Placebo Comparator): Multiple dose administration of Placebo (matching VNRX-5133 + VNRX-5022)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VNRX-5133 — β-lactamase inhibitor
  Arms: Part 1A; Part 1B; Part 2 - 2A; Part 2 - 2B
Drug: VNRX-5022 — Approved β-lactam antibiotic
  Arms: Part 1A; Part 1B; Part 2 - 2A; Part 2 - 2B
Drug: Metronidazole — Approved antibiotic and antiprotozoal medication
  Arms: Part 1B
Drug: Placebo — Placebo (matching VNRX-5133 + VNRX-5022)
  Arms: Part 2 - 2C

SUMMARY:
This is a 2-part, drug-drug interaction study to evaluate potential PK interactions after single doses in Part 1 and multiple doses in Part 2. In Part 1, subjects will receive single dose of 5 treatments in a cross-over design; in Part 2 subjects will receive treatment for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Males or non-pregnant, non-lactating females
* Body Mass Index (BMI) between 18.5 - 32.0, inclusive
* Weight greater than or equal to 50 kg
* Suitable veins for cannulation

Exclusion Criteria:

* Employee of site or the sponsor
* Any disease that poses an unacceptable risk to participants
* Abnormal ECG
* Abnormal labs
* Abnormal vital signs
* Current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorder
* Positive serology for hepatitis B surface antigen, hepatitis C antibody, or human immunodeficiency virus (HIV) type 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) of VNRX-5133 and VNRX-5022 following single doses alone and in combination (Part 1A) | 0-48 hours
  Cmax
Area under the plasma concentration versus time curve (AUC) of VNRX-5133 and VNRX-5022 following single doses alone and in combination (Part 1A) | 0-48 hours
  AUCinf

SECONDARY OUTCOMES:
Peak Plasma Concentration (Cmax) of metronidazole, VNRX-5133, and VNRX-5022 (Part 1B) | 0-48 hours
  Cmax
Area under the plasma concentration versus time curve (AUC) of metronidazole, VNRX-5133, and VNRX-5022 (Part 1B) | 0-48 hours
  AUCinf
Number of Subjects with Treatment Emergent Adverse Events | First dose to 7 days after last dose: Part 1: 20 days / Part 2: 17 days
  TEAEs based on patient reporting, physical exams, collection of vital signs, ECGs and absolute values and changes over time of hematology, chemistry and urinalysis.
Accumulation of VNRX-5133 + VNRX-5022 following multiple dose administration | Part 2: 10 days
  Trough concentration levels from Day 1 - Day 10

OTHER OUTCOMES:
Bactericidal titers (Part 2) | 10 days
  To evaluate serum and urine bactericidal activity at peak and trough concentrations following multiple dose administration of VNRX-5133 + VNRX-5022

CONTACTS AND LOCATIONS:
Locations (1):
- PRAHS, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: No